CLINICAL TRIAL: NCT06612983
Title: Effects of Instrument Assisted Soft Tissue Mobilization on Healthy Tissue Regarding Range of Motion and Gait
Acronym: (IASTM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Marschner (Other)
Collaborators: Minot State University (Other)
Responsible Party: Sponsor-Investigator, Beth Marschner, Assistant Professor, Minot State University
Organization: Minot State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2242
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Instrument assisted soft tissue mobilization; Range of Motion; Gait

STUDY DESIGN:
Intervention Model Description: All participants will experience the IASTM treatment first and the first session and the walking - sham treatment at the second session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IASTM (Experimental): This arm of the study received treatment on day one and walking treatment on day two.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization; Other: Walking Treatment

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — Instrument assisted soft tissue mobilization is a technique that is applied using specially designed tools/instruments to provide a mobilizing effect to soft tissues including the skin, fascia, muscles, and tendons by its various direct compressive stroke techniques on the gastroc/soleus complexes and Achilles tendons in the first session.
  Other Names: HawkGrips
Other: Walking Treatment — Movement itself should promote mobility so walking steadily for the same period of time as the IASTM had taken to complete is the sham treatment in second session.

SUMMARY:
The goal of this clinical trial is to study the effects of instrument assisted soft tissue mobilization (IASTM) in healthy tissue of adult volunteers. The main questions it aims to answer are:

* Does IASTM treatment have an effect on range of motion (ROM) as measured in the ankle and knee?
* Does IASTM treatment have an effect on movement patterns including gait - how a person walks? Researchers will compare pre-test and post-test data from the same individual on their day with treatment to the pre-test and post-test data from the same individual on their day without treatment to see if ROM or gait are effected by use of IASTM.

Participants will:

* Complete a past medical and injury history questionnaire
* Have ankle and knee range of motion (ROM) measurements taken on both lower extremities using a goniometer
* Undergo a gait analysis to determine center of gravity, center of pressure, step length, stride length, and stride frequency using Noraxon MyoMuscle Ultium Insoles
* Undergo IASTM treatment techniques using the HawkGrips tools including applying emollient to the skin to reduce friction on the surface followed by scanning the gastroc/soleus complexes and Achilles tendons using the HG8-Scanner tool for 15 strokes in each direction to identify areas of concern, then the concave tool corresponding to the size of the structure being treated will be used (HG6-Large Multi-Curve, HG5-Medium Multi-Curve, HG4-Small Multi-Curve) for 15 strokes in each direction. Treatment techniques should last for 10 minutes in total on each side.
* Complete the ankle and knee ROM measurements as well as gait analysis again to document progress at the end of the first session.
* Return three to seven days after the first session in which the subject will have the walking treatment.
* Undergo the same baseline pre-test measurements for range of motion and gait analysis as the first session
* Experience the walking treatment by walking for the same time period that the IASTM treatment took at the first session
* Undergo the post-test range of motion and gait analysis for data comparison.

DETAILED DESCRIPTION:
No further information to note than what is described in the summary or elsewhere

ELIGIBILITY:
Inclusion Criteria:

* Individuals from a small regional university student body, faculty and staff may choose to volunteer to participate in this study.

Exclusion Criteria:

* Acute spinal cord injury with neurological deficits
* Neurological disorders
* Acute lower extremity injury such as sprain or strain
* Acute lower extremity pain causing gait deviation
* Any type of lower extremity fracture within the past 12 months
* Lumbar disc pathology with radicular symptoms
* Use of blood thinning or clotting medications
* Known connective tissue disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Range of Motion | From baseline to end of session at one hour
  Bilateral knee flexion and extension as well as ankle plantarflexion, dorsiflexion, inversion and eversion range of motion measurements were taken in supine using a goniometer.
Gait | From baseline to end of session at one hour
  Gait analysis was conducted using Noraxon MyoMuscle System with Ultium insoles placed in the participants shoes. The software collected data on center of gravity, center of pressure, step length, stride length, and stride frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Marschner, DPT, Principal Investigator — Minot State University
Locations (1):
- Minot State University, Minot, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data is not the main focus of this study. The overall findings of the study with the larger number of participants to look at the trend is what will be shared (presented or published). The IRB proposal for this study included confidentiality of each individual participant as that will be maintained, but the global findings are what will be shared after data analysis for comparison.